CLINICAL TRIAL: NCT03927092
Title: Reliability and Validity of the Turkish Version of the Multiple Sclerosis Knowledge Questionnaire
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, Ece Cinar, Principal investigator, Ege University
Other Study IDs: 16-4.1/19
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; surveys and questionnaires; diagnostic self evaluation
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Multiple Sclerosis patients: Patients that attended an annual patient education seminar at the investigators' university hospital were asked to fill out the Turkish version of the Multiple Sclerosis Knowledge Questionnaire
  Interventions: Other: Multiple Sclerosis Knowledge Questionnaire

INTERVENTIONS:
Other: Multiple Sclerosis Knowledge Questionnaire — A 25-item self-administered questionnaire

SUMMARY:
Multiple Sclerosis Knowledge Questionnaire (MSKQ) is a 25-item self administered questionnaire assessing a patient's level of knowledge regarding multiple sclerosis (MS). Turkish translation of the questionnaire was prepared and participants in the annual patient education seminar in the investigators' university hospital were asked to answer these questions before and after the seminar.Their results were analysed to assess their level of knowledge about their disease.

DETAILED DESCRIPTION:
Multiple sclerosis knowledge questionnaire was developed in Italy (1) and was reported to be useful in measuring patients' level of knowledge about their disease. The English version of the questionnaire was translated into Turkish by three physicians than back translated into English by two separate linguists. Initially 5 MS patients were asked to answer this first version of the questionnaire and report any difficulties in understanding the items. Their feedback was used to give the questionnaire its final shape. For the validation stage, patients that were diagnosed as having MS and who attended the annual MS patient education seminar were enrolled into the study. They answered the questions twice, before and after the seminar. Their answers were analysed to measure their level of knowledge about their disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having Multiple Sclerosis
* Attends the annual patient education seminar at the investigators' university hospital
* Older than 18 years of age
* Can read and write

Exclusion Criteria:

* Does not accept to answer the questionnaire
* Unable to answer the questions due to a cognitive impairment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed as having multiple sclerosis.
Sampling Method: Non-Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
reliability of the questionnaire | 1 day
  Internal consistency was evaluated by the coefficient alpha (α) or Cronbach's coefficient, and if the Cronbach's coefficient value was greater than 0.7, it was considered as an acceptable internal consistency

SECONDARY OUTCOMES:
Number of correct answers | 1 day
  To assess the distribution of correct and false answers and the levels of significance, Chi-square test was used. To compare the two questionnaires answered by the same patient before and after the seminar Wilcoxon signed-rank test was used.

CONTACTS AND LOCATIONS:
Overall Officials: Ece Cinar, M.D., Principal Investigator — Ege University School of Medicine; Yesim Akkoc, M.D., Study Director — Ege University School of Medicine; Funda Calis, M.D., Principal Investigator — Ege University School of Medicine; Musa Baklaci, M.D., Principal Investigator — Ege University School of Medicine; Ozgul Ekmekci, M.D., Principal Investigator — Ege University School of Medicine; Ayse N Yuceyar, M.D., Principal Investigator — Ege University School of Medicine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giordano A, Uccelli MM, Pucci E, Martinelli V, Borreani C, Lugaresi A, Trojano M, Granella F, Confalonieri P, Radice D, Solari A; SIMS-Trial group. The Multiple Sclerosis Knowledge Questionnaire: a self-administered instrument for recently diagnosed patients. Mult Scler. 2010 Jan;16(1):100-11. doi: 10.1177/1352458509352865. Epub 2009 Dec 7. PMID 19995834